CLINICAL TRIAL: NCT07174687
Title: Efficacy of Dapagliflozin in the Progression of Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: SGLT2 Inhibitors in Geographic Atrophy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rajendra S. Apte, Principal Investigator; Paul A. Cibis Distinguished Professor of Ophthalmology and Visual Sciences; Vice Chair for Innovation and Translation, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202507116
Record Dates: First submitted 2025-09-05; First posted 2025-09-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Retinal Degeneration; Retinal Diseases; Eye Diseases; Geographic Atrophy; Pathological Conditions, Anatomical
Keywords: Geographic Atrophy (GA); Age-related Macular Degeneration; AMD; SGLT2; Dapagliflozin
MeSH Terms: conditions — Retinal Degeneration; Retinal Diseases; Eye Diseases; Geographic Atrophy; Pathological Conditions, Anatomical; Macular Degeneration | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either dapagliflozin or placebo and followed concurrently for 12 months. Two arms are defined: Experimental (Dapagliflozin 10 mg PO daily) and Placebo Comparator (matching placebo PO daily), with identical visit schedules for imaging and safety monitoring.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10 mg daily for 12 months (Experimental): Dapagliflozin 10 mg daily PO for 12 consecutive months
  Interventions: Drug: Dapagliflozin
- Matching Placebo for 12 months (Placebo Comparator): Subjects will receive a placebo medication daily PO for 12 consecutive months
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin is an SGLT2 inhibitor used in diabetes, heart failure, and chronic kidney disease patients.
  Other Names: Farxiga
  Arms: Dapagliflozin 10 mg daily for 12 months
Other: Matching Placebo — Matching oral placebo to dapagliflozin
  Arms: Matching Placebo for 12 months

SUMMARY:
AMD is a leading cause of blindness in individuals over 50 years old, with dry AMD being the most common form. Geographic atrophy (GA) is an advanced stage of dry AMD characterized by progressive retinal cell degeneration. The primary objectives of the study are to assess the safety, tolerability, and evidence of activity of SGLT2 inhibitors in subjects with Geographic Atrophy associated with AMD.

DETAILED DESCRIPTION:
This is a Phase II, prospective, single-center, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, and efficacy of oral dapagliflozin in subjects with geographic atrophy (GA) secondary to age-related macular degeneration (AMD).

The study will randomize approximately 70 subjects to obtain at least 60 evaluable subjects at a single center site.

Subjects will be randomized in a 1:1 manner to receive:

1. Dapagliflozin 10 mg (oral) once daily
2. Matching placebo (oral) once daily

Primary outcome of interest will be progression of GA lesion area over the 1-year period measured by fundus autofluorescence (FAF) , and secondary outcomes include structural and functional testing for visual function such as change in drusen volume as measured by OCT, dark adaptation, and low luminance BCVA to determine the effect of dapagliflozin on the progression of dry AMD.

All subjects will return for a final follow-up visit at Month 12, marking the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol
2. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
3. Participant is male or, if female, participant is surgically sterilized or amenorrheic for at least one year
4. ≥50 years old
5. Evidence of dry advanced AMD with the presence of non-foveal Geographic Atrophy (GA)

   1. The geographic atrophy must not involve the center point of the fovea.
   2. Total area of geographic atrophy must be between 2.5 mm2 and 17.5 mm2 (1 - 4 disc areas, respectively).
   3. If the geographic atrophy consists of multiple lesions, at least one lesion must have an area of ≥1.25 mm² (equivalent to 0.5 disc areas).
6. BCVA between 20/25 and 20/320
7. Must be treatment-naïve for AMD, except for oral supplements

Exclusion Criteria:

1. Prior investigational drug use within 60 days
2. Use of other SGLT2 inhibitors
3. History of symptomatic hypotension or symptomatic hypotension (symptoms of hypotension + SBP < 90mmHg) at baseline
4. Type I and Type II Diabetes Mellitus
5. End stage renal disease or estimated glomerular filtration rate less than 25 mL/min/1.73 m2 per MDRD calculation
6. History of heart failure
7. History of a serious hypersensitivity reaction to dapagliflozin or any of the excipients in FARXIGA
8. Other concomitant disease or condition that investigator deems unsuitable for the study, including drug or alcohol abuse or psychiatric, behavioral, or cognitive disorders, sufficient to interfere with the patient's ability to understand and comply with the study instructions or follow-up procedures
9. Any prior treatment for AMD (dry or wet) or any prior intravitreal treatment for any indication in either eye, except oral supplements of vitamins or mineral
10. Any intraocular surgery or thermal laser within 3 months of date of randomization
11. Any ocular or periocular infection (including blepharitis), or ocular surface inflammation in the past 12 weeks
12. Any prior thermal laser in the macular region, regardless of indication (self-report)
13. Any evidence of choroidal neovascularization in study eye
14. Enrollment in another interventional trial during the trial period

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in Square Root GA Lesion Size in the Study Eye at Month 12 | Baseline (screening) and Month 12.
  The square root GA lesion size (i.e. transformed area of GA) was measured by FAF photographs at baseline and 12 months. Baseline is defined as the last available, non-missing observation prior to first study drug administration.

SECONDARY OUTCOMES:
Mean Change From Baseline in Drusen Size in the Study Eye at Month 12 | Baseline (screening) and Month 12.
  The mean change in size of drusen volume measured by OCT from Baseline to Month 12
Mean Change From Baseline in best corrected visual acuity (ETDRS letters) from Baseline to Month 12 | Baseline (screening) and Month 12.
  The mean change in best corrected visual acuity (ETDRS letters) from Baseline to Month 12
Mean Change From Baseline in Dark Adaptation in the Study Eye at Month 12 | Baseline (screening) and Month 12.
  The mean change in rod intercept time on dark adaptation from Baseline to Month 12
Mean Change From Baseline in low luminance best corrected visual acuity (ETDRS letters) from Baseline to Month 12 | Baseline (screening) and Month 12.
  The mean change in low luminance best corrected visual acuity (ETDRS letters) from Baseline to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra S Apte, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the study team due to the small sample size and the associated risk of re-identification in this single-site pilot trial. In place of IPD sharing, de-identified, aggregate results will be disseminated through peer-reviewed publications and presentations, and summary-level data may be made available upon reasonable request.

REFERENCES:
- [Background] Yao S, Zheng F, Yu Y, Zhan Y, Xu N, Luo G, Zheng L. Apolipoprotein M promotes cholesterol uptake and efflux from mouse macrophages. FEBS Open Bio. 2021 Jun;11(6):1607-1620. doi: 10.1002/2211-5463.13157. Epub 2021 May 2. PMID 33830664
- [Background] Wolfrum C, Poy MN, Stoffel M. Apolipoprotein M is required for prebeta-HDL formation and cholesterol efflux to HDL and protects against atherosclerosis. Nat Med. 2005 Apr;11(4):418-22. doi: 10.1038/nm1211. Epub 2005 Mar 27. PMID 15793583
- [Background] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Background] Sunness JS, Gonzalez-Baron J, Applegate CA, Bressler NM, Tian Y, Hawkins B, Barron Y, Bergman A. Enlargement of atrophy and visual acuity loss in the geographic atrophy form of age-related macular degeneration. Ophthalmology. 1999 Sep;106(9):1768-79. doi: 10.1016/S0161-6420(99)90340-8. PMID 10485549
- [Background] Solini A, Giannini L, Seghieri M, Vitolo E, Taddei S, Ghiadoni L, Bruno RM. Dapagliflozin acutely improves endothelial dysfunction, reduces aortic stiffness and renal resistive index in type 2 diabetic patients: a pilot study. Cardiovasc Diabetol. 2017 Oct 23;16(1):138. doi: 10.1186/s12933-017-0621-8. PMID 29061124
- [Background] Schatz H, McDonald HR. Atrophic macular degeneration. Rate of spread of geographic atrophy and visual loss. Ophthalmology. 1989 Oct;96(10):1541-51. doi: 10.1016/s0161-6420(89)32694-7. PMID 2587050
- [Background] Sarks JP, Sarks SH, Killingsworth MC. Evolution of geographic atrophy of the retinal pigment epithelium. Eye (Lond). 1988;2 ( Pt 5):552-77. doi: 10.1038/eye.1988.106. PMID 2476333
- [Background] Ruiz M, Okada H, Dahlback B. HDL-associated ApoM is anti-apoptotic by delivering sphingosine 1-phosphate to S1P1 & S1P3 receptors on vascular endothelium. Lipids Health Dis. 2017 Feb 8;16(1):36. doi: 10.1186/s12944-017-0429-2. PMID 28179022
- [Background] Potter JW, Thallemer JM. Geographic atrophy of the retinal pigment epithelium: diagnosis and vision rehabilitation. J Am Optom Assoc. 1981 Jun;52(6):503-8. PMID 7264141
- [Background] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Maguire P, Vine AK. Geographic atrophy of the retinal pigment epithelium. Am J Ophthalmol. 1986 Nov 15;102(5):621-5. doi: 10.1016/0002-9394(86)90535-0. PMID 3777083
- [Background] Maayah ZH, Ferdaoussi M, Takahara S, Soni S, Dyck JRB. Empagliflozin suppresses inflammation and protects against acute septic renal injury. Inflammopharmacology. 2021 Feb;29(1):269-279. doi: 10.1007/s10787-020-00732-4. Epub 2020 Jun 20. PMID 32564182
- [Background] Leibowitz HM, Krueger DE, Maunder LR, Milton RC, Kini MM, Kahn HA, Nickerson RJ, Pool J, Colton TL, Ganley JP, Loewenstein JI, Dawber TR. The Framingham Eye Study monograph: An ophthalmological and epidemiological study of cataract, glaucoma, diabetic retinopathy, macular degeneration, and visual acuity in a general population of 2631 adults, 1973-1975. Surv Ophthalmol. 1980 May-Jun;24(Suppl):335-610. PMID 7444756
- [Background] Lambers Heerspink HJ, de Zeeuw D, Wie L, Leslie B, List J. Dapagliflozin a glucose-regulating drug with diuretic properties in subjects with type 2 diabetes. Diabetes Obes Metab. 2013 Sep;15(9):853-62. doi: 10.1111/dom.12127. Epub 2013 Jun 5. PMID 23668478
- [Background] Kosiborod M, Gause-Nilsson I, Xu J, Sonesson C, Johnsson E. Efficacy and safety of dapagliflozin in patients with type 2 diabetes and concomitant heart failure. J Diabetes Complications. 2017 Jul;31(7):1215-1221. doi: 10.1016/j.jdiacomp.2017.02.001. Epub 2017 Feb 10. PMID 28284707
- [Background] Kohler S, Zeller C, Iliev H, Kaspers S. Safety and Tolerability of Empagliflozin in Patients with Type 2 Diabetes: Pooled Analysis of Phase I-III Clinical Trials. Adv Ther. 2017 Jul;34(7):1707-1726. doi: 10.1007/s12325-017-0573-0. Epub 2017 Jun 19. PMID 28631216
- [Background] Kim SR, Lee SG, Kim SH, Kim JH, Choi E, Cho W, Rim JH, Hwang I, Lee CJ, Lee M, Oh CM, Jeon JY, Gee HY, Kim JH, Lee BW, Kang ES, Cha BS, Lee MS, Yu JW, Cho JW, Kim JS, Lee YH. SGLT2 inhibition modulates NLRP3 inflammasome activity via ketones and insulin in diabetes with cardiovascular disease. Nat Commun. 2020 May 1;11(1):2127. doi: 10.1038/s41467-020-15983-6. PMID 32358544
- [Background] Holz FG, Strauss EC, Schmitz-Valckenberg S, van Lookeren Campagne M. Geographic atrophy: clinical features and potential therapeutic approaches. Ophthalmology. 2014 May;121(5):1079-91. doi: 10.1016/j.ophtha.2013.11.023. Epub 2014 Jan 14. PMID 24433969
- [Background] Guo Z, Javaheri A. Empagliflozin to Prevent Doxorubicin Cardiotoxicity. JACC CardioOncol. 2025 Feb;7(2):185-187. doi: 10.1016/j.jaccao.2025.01.005. PMID 39967205
- [Background] Guo Z, Valenzuela Ripoll C, Picataggi A, Rawnsley DR, Ozcan M, Chirinos JA, Chendamarai E, Girardi A, Riehl T, Evie H, Diab A, Kovacs A, Hyrc K, Ma X, Asnani A, Shewale SV, Scherrer-Crosbie M, Cowart LA, Parks JS, Zhao L, Gordon D, Ramirez-Valle F, Margulies KB, Cappola TP, Desai AA, Pedersen LN, Bergom C, Stitziel NO, Rettig MP, DiPersio JF, Hajny S, Christoffersen C, Diwan A, Javaheri A. Apolipoprotein M Attenuates Anthracycline Cardiotoxicity and Lysosomal Injury. JACC Basic Transl Sci. 2023 Jan 4;8(3):340-355. doi: 10.1016/j.jacbts.2022.09.010. eCollection 2023 Mar. PMID 37034289
- [Background] Dudka LT, Inglis HJ, Johnson RE, Pechinski JM, Plowman S. Inequality of inspired and expired gaseous nitrogen in man. Nature. 1971 Jul 23;232(5308):265-8. doi: 10.1038/232265b0. No abstract available. PMID 4937081
- [Background] Ghanim H, Abuaysheh S, Hejna J, Green K, Batra M, Makdissi A, Chaudhuri A, Dandona P. Dapagliflozin Suppresses Hepcidin And Increases Erythropoiesis. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgaa057. doi: 10.1210/clinem/dgaa057. PMID 32044999
- [Background] Feuer WJ, Yehoshua Z, Gregori G, Penha FM, Chew EY, Ferris FL, Clemons TE, Lindblad AS, Rosenfeld PJ. Square root transformation of geographic atrophy area measurements to eliminate dependence of growth rates on baseline lesion measurements: a reanalysis of age-related eye disease study report no. 26. JAMA Ophthalmol. 2013 Jan;131(1):110-1. doi: 10.1001/jamaophthalmol.2013.572. No abstract available. PMID 23307222
- [Background] Elsoe S, Ahnstrom J, Christoffersen C, Hoofnagle AN, Plomgaard P, Heinecke JW, Binder CJ, Bjorkbacka H, Dahlback B, Nielsen LB. Apolipoprotein M binds oxidized phospholipids and increases the antioxidant effect of HDL. Atherosclerosis. 2012 Mar;221(1):91-7. doi: 10.1016/j.atherosclerosis.2011.11.031. Epub 2011 Nov 27. PMID 22204862
- [Background] Christoffersen C, Obinata H, Kumaraswamy SB, Galvani S, Ahnstrom J, Sevvana M, Egerer-Sieber C, Muller YA, Hla T, Nielsen LB, Dahlback B. Endothelium-protective sphingosine-1-phosphate provided by HDL-associated apolipoprotein M. Proc Natl Acad Sci U S A. 2011 Jun 7;108(23):9613-8. doi: 10.1073/pnas.1103187108. Epub 2011 May 23. PMID 21606363
- [Background] Christoffersen C, Jauhiainen M, Moser M, Porse B, Ehnholm C, Boesl M, Dahlback B, Nielsen LB. Effect of apolipoprotein M on high density lipoprotein metabolism and atherosclerosis in low density lipoprotein receptor knock-out mice. J Biol Chem. 2008 Jan 25;283(4):1839-47. doi: 10.1074/jbc.M704576200. Epub 2007 Nov 15. PMID 18006500
- [Background] Christensen PM, Liu CH, Swendeman SL, Obinata H, Qvortrup K, Nielsen LB, Hla T, Di Lorenzo A, Christoffersen C. Impaired endothelial barrier function in apolipoprotein M-deficient mice is dependent on sphingosine-1-phosphate receptor 1. FASEB J. 2016 Jun;30(6):2351-9. doi: 10.1096/fj.201500064. Epub 2016 Mar 8. PMID 26956418
- [Background] Bonnet F, Scheen AJ. Effects of SGLT2 inhibitors on systemic and tissue low-grade inflammation: The potential contribution to diabetes complications and cardiovascular disease. Diabetes Metab. 2018 Dec;44(6):457-464. doi: 10.1016/j.diabet.2018.09.005. Epub 2018 Sep 26. PMID 30266577
- [Background] Apte RS. Age-Related Macular Degeneration. N Engl J Med. 2021 Aug 5;385(6):539-547. doi: 10.1056/NEJMcp2102061. PMID 34347954
- [Background] Demaria R, Picard E, Bodino M, Aymard T, Albat B, Frapier JM, Chaptal PA. [Migration of a clavicular bone wire acutely perforating the ascending aorta]. Presse Med. 1998 Jun 13;27(21):1013. No abstract available. French. PMID 9767821

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT07174687/Prot_SAP_000.pdf